CLINICAL TRIAL: NCT04219345
Title: Transcranial Direct Current Stimulation Associated With Mindfulness in Chronic Migraine: a Randomized Clinical Trial
Brief Title: Transcranial Direct Current Stimulation Associated With Mindfulness in Chronic Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Ph.D, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Mindfulness/ tDCS in migraine
Record Dates: First submitted 2019-09-16; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, placebo-controlled clinical trial will analyze patients with a confirmed diagnosis of chronic migraine by a neurologist who were subjected to tDCS associated with mindfulness practices.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): In the group A will be administered anodic tDCS and instructed in mindfulness practices.
  Interventions: Device: Transcranial direct current stimulation
- Sham group (Sham Comparator): In the group B will be administered sham tDCS and instructed in mindfulness practices.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Both groups will undergo the same protocol of twelve sessions of twenty minutes of tDCS associated with mindfulness, where only the type of received electric current is varied (active or simulated sham type). The twelve sessions will be performed in three sessions per week for four weeks, and mindfulness practice at home will be encouraged on days when the intervention is not administered.
  Other Names: Mindfulness

SUMMARY:
This study is a group controlled clinical trial. ParallelParallel study, patients aged 25-50 years, with Migraine Chronicle. Twelve sessions will be held during four mindfulness practice with four recordings (one per week). As a brainwave biomarker, the Muse, a Electroencephalogram (EEG). The investigators will use the MIDAS questionnaire, the HIT-6 Questionnaire and the FFMQ-BR. Based on the use of tDCS in patients with chronic pain, and in benefits of Mindfulness practice in these patients, the objective is to evaluate if the mindfulness-associated TCCA provides satisfactory results in the painful prophylaxis of patients with chronic migraine.

DETAILED DESCRIPTION:
Background: Chronic Migraine is a difficult to diagnose disease whose symptoms affect the quality of life of those affected. This study is a group controlled clinical trial. ParallelParallel study, patients aged 25-50 years, with Migraine Chronicle Methods / Design: Will be held at the Aging Studies Laboratory and Neuroscience of the Federal University of Paraíba. Twelve sessions will be held during four mindfulness practice with four recordings (one per week). As a brainwave biomarker, the Muse, a Electroencephalogram (EEG). The investigators will use the MIDAS questionnaire Migraine Disability), the HIT-6 Questionnaire (Headache Impact Test) and the FFMQ-BR (Five Facet Mindfulness Questionnaire). The investigators will analyze the data through Statistical Package for Social Sciences (SPSS) 25.0 program for software and from data normality analysis will be applied parametric and / or nonparametric tests.

Discussion: Based on the use of tDCS in patients with chronic pain, and in benefits of Mindfulness practice in these patients, the objective is to evaluate if the mindfulness-associated TCCA provides satisfactory results in the painful prophylaxis of patients with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged between twenty-five and fifty years who have been clinically diagnosed with chronic migraine according to the third edition of the International Classification of Headache Disorders (ICHD-3) will be selected.
* Only patients who are able to complete treatment in the twelve sessions of four preprogrammed consecutive weeks will be accepted, although up to three alternating absences or two excused absences are tolerated.
* Absent days will be replaced with follow-up on the next working day to minimize dropouts and promote adherence to treatment. Flextime will be provided to participants who receive the therapy, as well as direct contact by calling participants by phone to confirm the evaluation dates and reinforce adherence to treatment.

Exclusion Criteria:

* Exclusion criteria will be the presence of headache attributed to another neurological or associated neuropsychiatric pathology, the use of central nervous system (CNS)-modulating drugs, the diagnosis of a severe, distinct neurological or psychiatric disease, the use of another nondrug therapy for migraine or other CNS pathologies concurrent with or immediately before the intervention, the presence of metallic implants located in the cephalic region and the implantation of cardiac pacemakers.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Migraine disabIlity assessment questionnaire - MIDAS | 04 weeks
  The Migraine Disability Assessment Questionnaire (MIDAS) will be used for this assessment. Its objective is to evaluate the inability of migraine patients to perform daily and professional tasks. This instrument contains five questions that must be completed with the number of days the patient failed to perform the specified activity because he or she was experiencing a migraine episode. This assessment is a useful tool for identifying the severity of this condition. Includes questions that score between 8 and 13 points, depending on the answer given. This questionnaire can be applied to people of different educational and social levels, as it is considered easy to answer (FRAGOSO, 2002).

SECONDARY OUTCOMES:
Headache impact test - HIT-6 | 04 weeks
  HIT-6 is a highly reliable questionnaire validated in Portuguese. It evaluates the frequency of headache impact on the quality of life of patients with chronic and episodic migraine and discriminates the types of migraine presented by the patient (episodic, chronic or non-migratory types). It is simple and easy to apply (Yang et al, 2010). This questionnaire consists of six questions that evaluate these parameters through the following options: never, rarely, sometimes, very often and always. A predetermined value is associated with each of these frequency parameters (for example, the score is rarely 8 points and usually 13 points), which will be added to the final score to determine the score equivalent to the headache impact.
Five facets of mindfulness questionnaire (FFMQ-BR) | 04 weeks
  The FFMQ-BR is an instrument for assessing the characteristics of mindfulness validated in Brazil in 2014. Subdivided into five main evaluation factors (observation, description, non-judgment, non-reactivity and conscientious acting) assessed in the situations addressed in each item - For example, "In difficult situations, I can pause without reacting immediately." This scenario is classified by the participant through a scale ranging from 1 to 5 points, where 1 represents "never or almost never" and 5 represents "always or almost always" (BARROS et al, 2014). The total score of the questionnaire will be calculated and this score will be compared before and after all intervention sessions are completed between the two groups to assess whether the participants' level of attention has increased.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraíba
Locations (2):
- Brazil (2):
  - Suellen Marinho Andrade, João Pessoa, Paraíba
  - Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba

IPD SHARING:
Plan to Share IPD: No